CLINICAL TRIAL: NCT03542734
Title: The Associations of Retinal Microvascular Signs and Brain Imaging Markers With Cognitive Impairment in Patients With Small Vessel Disease
Brief Title: Cognitive Impairment, Retinopathy, and Cerebrovascular Lesions in the Elderly
Acronym: CIRCLE
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: CIRCLE-CHINA
Record Dates: First submitted 2018-05-20; First posted 2018-05-31 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Small Vessel Diseases; Retinopathy; Cognitive Dysfunction
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Retinal Diseases; Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with SVDs: Individuals with at least one following imaging finding: recent small subcortical infarcts, lacunes, white matter hyperintensities, perivascular spaces, microbleeds, or brain atrophy on baseline brain MRI.
  Interventions: Other: multimodal magnetic resonance imaging
- Individuals without SVDs: Individuals without any following imaging finding: recent small subcortical infarcts, lacunes, white matter hyperintensities, perivascular spaces, microbleeds, or brain atrophy on baseline brain MRI.
  Interventions: Other: multimodal magnetic resonance imaging

INTERVENTIONS:
Other: multimodal magnetic resonance imaging — multimodal magnetic resonance imaging included T1, FLAIR, MRA, PWI and/or ASL, DTI, DKI, SWI, fMRI
  Other Names: retinal digital images; neuropsychological testing; Blood samples collection

SUMMARY:
The CIRCLE study is a single-center prospective observational study that enrolled individuals with cerebral small vessel disease (SVD), while free of known dementia or stroke (both cerebral infarction and hemorrhage). The patients will receive neuropsychological testing, retinal digital images and multimodal magnetic resonance imaging (MRI). Blood samples will also be collected. Recent small subcortical infarcts, lacunes, white matter hyperintensities, perivascular spaces, microbleeds, and brain atrophy will be evaluated on both baseline and follow-up brain MRIs. The investigators will explore the predictors of preogression of SVD and cognitive deficits.

DETAILED DESCRIPTION:
Cerebral small vessel disease (SVD) is commonly detected in elderly individuals, and patients with stroke or neurodegenerative disease. Features seen on neuroimaging include recent small subcortical infarcts, lacunes, white matter hyperintensities, perivascular spaces, microbleeds, and brain atrophy. Previous studies indicated that SVD was associated with an increased risk of stroke and stroke recurrence, cognitive deficits, physical disabilities, and mortality. However the pathogenesis of SVD is largely unknown. Little is known about how SVD lesions contribute to neurological or cognitive symptoms, and the association with risk factors. Recent data sugessted concomitant SVDs and retinopathy is associated with a profile of vascular cognitive impairment. In this study, the investigators try to explore the new pathological mechanism of SVD, the new predictors for SVD progression, and the association with cognitive Impairment, based on digital retinal images and brain multimodal imaging technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥40y; no upper limit)
* Free of known dementia or stroke (both cerebral infarction and hemorrhage)

Exclusion Criteria:

* Any MRI contraindications
* Serious head injury (resulting to loss of consciousness) or received intracranial surgery
* Suffering from cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of certain towns
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive state | 1year
  Cognitive state based on Mini-mental State Examination

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen L, Zhong W, Chen H, Zhou Y, Ran W, He Y, Zhang T, Zhu X, Xu X, Yuan C, Lou M. ORIENT Diet: A Potential Neuroprotective Dietary Pattern for Chinese Stroke High-Risk Population. J Am Med Dir Assoc. 2025 Jan;26(1):105331. doi: 10.1016/j.jamda.2024.105331. Epub 2024 Oct 30. PMID 39488333
- [Derived] Lee DA, Lee HJ, Jo G, Park KM. Choroid plexus volumes in patients with transient global amnesia: A retrospective study. Medicine (Baltimore). 2024 Oct 11;103(41):e40077. doi: 10.1097/MD.0000000000040077. PMID 39465804
- [Derived] Zhao Y, Zhou Y, Zhou H, Gong X, Luo Z, Li J, Sun J, Lou M, Yan S. Low-density lipoprotein cholesterol, statin therapy, and cerebral microbleeds: The CIRCLE study. Neuroimage Clin. 2023;39:103502. doi: 10.1016/j.nicl.2023.103502. Epub 2023 Aug 22. PMID 37643520
- [Derived] Zhu X, Zhou Y, Zhong W, Li Y, Wang J, Chen Y, Zhang R, Sun J, Sun Y, Lou M. Higher Functional Connectivity of Ventral Attention and Visual Network to Maintain Cognitive Performance in White Matter Hyperintensity. Aging Dis. 2023 Aug 1;14(4):1472-1482. doi: 10.14336/AD.2022.1206. PMID 37163435
- [Derived] Zhang K, Zhou Y, Zhang W, Li Q, Sun J, Lou M. MRI-visible perivascular spaces in basal ganglia but not centrum semiovale or hippocampus were related to deep medullary veins changes. J Cereb Blood Flow Metab. 2022 Jan;42(1):136-144. doi: 10.1177/0271678X211038138. Epub 2021 Aug 25. PMID 34431378
- [Derived] Zhang W, Zhou Y, Wang J, Gong X, Chen Z, Zhang X, Cai J, Chen S, Fang L, Sun J, Lou M. Glymphatic clearance function in patients with cerebral small vessel disease. Neuroimage. 2021 Sep;238:118257. doi: 10.1016/j.neuroimage.2021.118257. Epub 2021 Jun 10. PMID 34118396